CLINICAL TRIAL: NCT03440125
Title: Cayenne Pepper Cataplasm Application and Potential Side Effects
Brief Title: Cayenne Pepper Cataplasm - Safety Study
Acronym: Munari04
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Primorska (Other)
Collaborators: S2P, Science to Practice, Ltd. (Other); Comenius University (Other); Wilhelminenspital Vienna (Other); Ludwig Boltzmann Institute of Electrical Stimulation and Physical Rehabilitation (Other)
Responsible Party: Principal Investigator, Nejc Sarabon, Dean of Faculty, University of Primorska
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UP-MunariStudy
Record Dates: First submitted 2018-02-06; First posted 2018-02-20 (Actual); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Capsicum; Physical Therapy; Pain
MeSH Terms: conditions — Low Back Pain; Pain | interventions — Electric Stimulation; Massage

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy (Experimental): Healthy participants with no low back pain. 20 min application of Cayenne Pepper Cataplasm (Cayenne Pepper topical) on the back will be administered.
  Interventions: Drug: Cayenne Pepper topical
- LBP patients - CPC Group (Experimental): Participants suffering from low back pain (LBP) receiving 10 times (within 3 weeks) 20min application of Cayenne Pepper Cataplasm (Cayenne Pepper topical).
  Interventions: Drug: Cayenne Pepper topical
- LBP patients - CPC and ES/M Group (Experimental): Participants suffering from low back pain (LBP) receiving 10 times (within 3 weeks) 20min application of Cayenne Pepper Cataplasm (Cayenne Pepper topical), and half of the subject also receiving 10 min electrical Stimulation and 10 min massage Treatment on the back.
  Interventions: Drug: Cayenne Pepper topical; Device: Electrical stimulation; Procedure: Massage

INTERVENTIONS:
Drug: Cayenne Pepper topical — 20min topical Cayenne Pepper Cataplasm application containing 5% Cayenne Pepper nd 95% Kaolin mixed with water
  Other Names: Cayenne Pepper Cataplasm application
Device: Electrical stimulation — Electrical stimulation 10min 60Hz biphasic rectangular neuromuscular electrical Stimulation (NMES)
  Other Names: Neuromuscular Electrical Stimulation (NMES)
  Arms: LBP patients - CPC and ES/M Group
Procedure: Massage — 10 minutes of classical massage of low back pain area.
  Other Names: Classical massage
  Arms: LBP patients - CPC and ES/M Group

SUMMARY:
The beneficial analgesic effects of Rubefacenciae (redden skin substances), is known since 1830 as a treatment for pain, cramps, and disorders of the musculoskeletal system. Herbal cataplasms containing rubefacient substances, such as Cayenne pepper, are commonly used as natural medications to treat painful or aching areas in the case of acute or chronic back pain, and rheumatisms. In Vienna and lower Austria, a Cayenne Pepper Cataplasm (CPC) application containing Cayenne pepper and Kaolin powder in mixed proportion, is commonly used to treat musculoskeletal conditions of pain especially of the low back. However, a concern about the safety of such applications was recently raised.

Therefore, the aims of the present study are to evaluate the effects of 10x 20min CP cataplasm application as a single treatment or in combination with electrical stimulation and massage on selected functional and molecular parameters on i) healthy subjects and ii) subjects suffering from low back pain.

DETAILED DESCRIPTION:
Musculoskeletal diseases, such as neck and low back pain, are widespread disorders in many developed countries. Their management is challenging, and it may have mounting socioeconomic burden. Several evidences in the literature demonstrate the efficacy of many therapeutic strategies in the treatment of these conditions, based on pharmacological or surgical interventions. Physical medicine therapies are good alternatives that may have beneficial effects, especially when used as first line of intervention before approaching more expensive pharmacological or invasive medications. The beneficial analgesic effects of Applicatio Epispasticorum of Rubefacenciae (redden skin substances), is known since 1830 as a treatment for pain, cramps, and disorders of the musculoskeletal system. Herbal cataplasms containing rubefacient substances, such as Cayenne pepper (CP), are commonly used as natural medications to treat painful or aching areas in the case of acute or chronic back pain, and rheumatisms. They are also used in pain involving joints caused by osteoarthritis. A galenic preparation composed of rubefacient substances of vegetable origin, which generated vasodilation and increase in blood circulation on the treated areas, was first prescribed in 1909 by Dr. Giuseppe Munari to treat pain of various areas of the locomotive system. He proposed a method based on applications prepared according to his own galenic formula that have become famous all over Italy and Europe. In Vienna and lower Austria, a Munari-like application containing CP and Kaolin powder in mixed proportion, is commonly used to treat musculoskeletal conditions of pain especially of the low back. The research on responses to CPC applications, particularly in combination with other modalities is scarce.

Therefore, the aims of the present study are firstly to evaluate the effects of 10x 20min CP cataplasm application on selected functional and molecular parameters on healthy subjects. Then, the same applications will be used on subjects suffering from low back pain (LBP) - both as a single treatment and in combination with electrical stimulation and massage.

ELIGIBILITY:
Inclusion Criteria:

* Chronic low back pain (>3 months)
* Body mass index below 35 kg/mˇ2

Exclusion Criteria:

* pregnancy
* sensibility disorders (e.g. due to neurological disease)
* injuries, open wounds or rash in intervention area
* known hypersensitivity against the applied substances
* HIV, Hepatitis C and other due blood communicable infectious diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-03-15 (Actual); Primary Completion 2016-11-15 (Actual); Study Completion 2016-12-15 (Actual)

PRIMARY OUTCOMES:
Change in concentration of circulating biomarkers of inflammation, neudroendocrine stress and blood vessel activation | Before the application, 45 minutes after 10th application and 48 hours after 10th application
  The blood analysis will include standard analysis of hemogram, C-reactive proteins, creatine-kinase, sedimentation, albumin and cortisol. Enzyme-linked immunosorbent assay (ELISA) will include Tumor necrosis factor-Alpha, Interleukin-6, Leukotriene B4 and P-Selectine. Additionally, microRNA analysis will be performed (gene numbers: 1, 21, 23, 25, 103, 126, 133, 146, 155, 199a, 199b, 191, 206, 451.
Change in systolic and diastolic blood pressure | Before the application, 45 minutes after 10th application and 48 hours after 10th application
  Systolic and diastolic blood pressure [mmHg], measured at both sides of the body with blood pressure gauge
Heart rate | Before the application, 45 minutes after 10th application and 48 hours after 10th application
  Heart rate (bpm), measured with heart rate monitor belt.

SECONDARY OUTCOMES:
36-Item Short Form Survey (SF-36) | Before the application, 45 minutes after 10th application and 48 hours after 10th application
  The Short Form (36) Health Survey (SF-36) is a patient-reported survey of patient health. It consists of eight scaled scores, which are the weighted sums all questions in their respective section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the higher is the disability.
Change in pain perception | Before the application, 45 minutes after 10th application and 48 hours after 10th application
  Pain perception during rest and movement assessed with visual analogue scale (0-10). 0 represents no pain, and 10 represents severe pain.
EQ-5D- 5L questionnaire | Before the application, 45 minutes after 10th application and 48 hours after 10th application
  EQ-5D- 5L questionnaire includes following aspects: mobility, care, usual activities, pain/discomfort, anxiety/depression, crosswalk-index, self-feeling of health. Each aspect is evaluated on a 1-5 scale, with following descriptions of levels: having no problems, having slight problems, having moderate problems, having severe problems and being unable to do/having extreme problems. Visual analogue scale is the second part of the questionnaire, asking to mark health status on the day of the interview on a 20 cm vertical scale with end points of 0 and 100. There are notes at the both ends of the scale that the bottom rate (0) corresponds to " the worst health you can imagine", and the highest rate (100) corresponds to "the best health you can imagine".
Oswestry disability index (ODI) | Before the application, 45 minutes after 10th application and 48 hours after 10th application
  ODI will be used only in LBP arms (Arm 2 and 3). ODI is commonly used by clinicians and researchers to quantify disability for low back pain.
Skin Sensory Function | Before the application, 45 minutes after 10th application and 48 hours after 10th application
  Skin sensory function will be assessed by 2-point discrimination test (which is carried out using two pins, oriented in medial-lateral direction and pressed perpendicularly to the skin, with the medial pin being 3 cm laterally from the L3 spinal process. The subject is asked to report whether he/she felt one or two pins) and mono filament/light touch sensitivity tests (monofilaments calibrated to 0.025, 0.07, 2, 5, and 10 grams The subject is asked to report when he/she felt touching the skin with a monofilament 3 cm laterally from L3 spinal process). The lightest mono filament and the lowest pin inter-distance are take as final outcome measures.
Flexibility | Before the application, 45 minutes after 10th application and 48 hours after 10th application
  Assessment of total spine flexibility (forward bend test) and separately for the lumbar part (Schober's test) and thoracic part.
Skin Temperature | Before the application, 45 minutes after 10th application and 48 hours after 10th application
  Skin temperature [°C] at the site of application (low back) and at the control part of the body (neck), measured with a laser thermometer.

CONTACTS AND LOCATIONS:
Overall Officials: Nejc Šarabon, PhD, Principal Investigator — Faculty of Health Sciences, University of Primorska, Slovenia
Locations (2):
- Facultiy of Physical Education and Sports, Comenius University of Bratislava, Bratislava, Slovakia
- Faculty of Health Sciences, Izola, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided